CLINICAL TRIAL: NCT06332924
Title: The Effect of Positive Birth Motivational Education on the Perception of Traumatic Birth in Primipara Pregnant Women
Brief Title: Primipara Pregnant Women and Motivational Interview
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Enzel Köksaldı, graduate student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/19
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: Positive birth; Motivational interviewing training; Primiparous pregnant women; Perception of traumatic birth
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: In the project, it was calculated that the experimental and control groups should have at least 30 observations each, and the sample of the study was calculated as 60 pregnant women. It was aimed to interview a total of 60 pregnant women, 30 in the control group and 30 in the experimental group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing group (Experimental): The patients in the intervention group will be informed about the study, and after the purpose and method of the study are explained, their consent will be obtained and the "Pregnant Information Form" will be applied.
  * There will be 3 meetings for both groups, one week apart. Interviews will include primipara pregnant women in their 30th, 32nd and 34th weeks of pregnancy.
  * Preliminary tests will be conducted before the interviews.
  * After the interviews are completed, final tests will be carried out and the study will be terminated.
  * Motivational Interviewing Training for the intervention group will be prepared in detail, with the aim of answering the pregnant woman's questions, and with methods that are relevant to her needs and interests by providing body awareness.
  Interventions: Behavioral: motivational discussion group
- Control group: (No Intervention): Scales will be applied to the control group as pre-test and post-test with a 2-week interval.

INTERVENTIONS:
Behavioral: motivational discussion group — There will be 3 interviews with the motivational interview group, one week apart.
  Other Names: control group
  Arms: Motivational interviewing group

SUMMARY:
The first birth is the most important moment a woman experiences in her life as she embarks on her motherhood journey. Waiting for the birth of a new life can be very exciting for mothers. Positive birth is an approach that asks the woman to approach her birth story from a positive perspective and to have a stronger, more impressive and positive birth experience. Primipara pregnant women especially benefit from and need this positive birth approach. Motivational interviews are interviews conducted to support positive births and to help women develop a positive attitude towards their birth experiences.

This planned study was planned as a randomized controlled trial with pre-test and post-test measurements, with the aim of determining the level of traumatic birth perception in primipara women who were given or not given training and examining the effects of positive birth motivational education by taking into account the need for education with numerical data.

ELIGIBILITY:
Inclusion Criteria:Must be between the ages of 20-35, have a primipara pregnancy (30-34 weeks of gestation), be a Turkish citizen, have no history of risky pregnancy, have no psychological disorders, and wish to participate in the study voluntarily.

-

Exclusion Criteria:Having an unplanned or involuntary pregnancy, having a threat of premature birth, wanting to leave the job at any time.

-

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Primipara Pregnant Women and Traumatic Birth | Once a week for 3 weeks
  motivational interviewing

CONTACTS AND LOCATIONS:
Overall Officials: enzel köksaldı, Study Director — SağlıkBilimleriU

IPD SHARING:
Plan to Share IPD: Undecided